CLINICAL TRIAL: NCT02358525
Title: Effects of a Multi-Modality Rehabilitation Program on Immune Activation, Depressive Symptoms and Quality of Life in Heart Failure Patients. A Pilot Study
Brief Title: Effects of a Rehabilitation Program on Immune Activation and Mood in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Ludwig-Boltzmann Institut fuer Rheumatologie, Balneologie und Rehabilitation (Other)
Responsible Party: Principal Investigator, Dr. Katherine Wachmann, Study coordinator, Ludwig-Boltzmann Institut fuer Rheumatologie, Balneologie und Rehabilitation
Other Study IDs: J3256
Record Dates: First submitted 2014-11-19; First posted 2015-02-09 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure; Depressive Symptoms
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: multi-modality rehabilitation program for heart failure — rehabilitation consists of supervised exercise training, both endurance and strength, as well as gymnastics, diet and psychosocial education around living with heart failure

SUMMARY:
The aim of this descriptive study is to examine potential changes regarding inflammatory cytokine levels, depressive symptoms and quality of life over the course of the 4-week inpatient rehabilitation program which includes a cassette of modalities including counseling, psychosocial education and supervised exercise training as a main pillar, and to further investigate if there are correlations between changes in immune regulation, depressive symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure with reduced ejection fraction (HFREF) with an EF ≤ 45%, NYHA (New York Heart Association) I - III; ACC/AHA (American College of Cariology/ American Heart Association) stage C, irrespective of etiology
* Clinically stable patients without deterioration or hospitalization due to heart failure within the last 4 weeks
* Neuro-hormonal medication according to the ESC (European Society of Cardiology) guidelines for the treatment of chronic heart failure consisting of antagonists of the Renin-Angiotensin-Aldosterone System (RAAS) and beta-blockers as indicated.
* Ability to fully understand all elements of and sign the written informed consent before initiation of the study

Exclusion Criteria:

* Fluid retention of cardiac decompensation, necessitating i.v. diuretic therapy
* Myocardial infarction within the last 2 months
* Surgery including cardiovascular or valvular surgery within 3 Months
* Uncontrolled proinflammatory comorbidities (e.g. Diabetes mellitus HbA1c >9%, COPD ( chronic obstructive pulmonary disease) >II, active rheumatic diseases and autoimmune disorders)
* Current infectious diseases ( e.g. pneumonia, COPD exacerbations or urinary tract infections)
* Morbid obesity: BMI > 40
* Alcohol or drug abuse
* psychiatric disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients, EF ≤ 45%, NYHA I - III; ACC/AHA stage C
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
inflammatory activity | 8 weeks
  levels of inflammatory biomarkers: Interleukin - 6, Tumor Necrosis Factor-alpha, Interleukin-1beta, Cellular Adhesion Molecule-1

SECONDARY OUTCOMES:
physical fitness | 8 weeks
  6-min-walk test
Quality of Life | 8 weeks
  questionnaires: SF-36 (short-form-36), KCCQ (Kansas City Cardiomyopathy Questionnaire), EQoL-5D (European Quality of LIfe-5Dimensions)
Depressive Symptoms | 8 weeks
  questionnaire: HADS (Hospital Anxiety and Depression Scale)

CONTACTS AND LOCATIONS:
Overall Officials: katherine wachmann, Dr., Principal Investigator — Ludwig Boltzmann IRBR
Locations (2):
- Austria (2):
  - Ska Rz Grossgmain, Grossgmain, Salzburg
  - SALK, 2.Medizin, HI-Ambulanz, Salzburg, Salzburg